CLINICAL TRIAL: NCT03307018
Title: Assessment of Influence of Routine Postoperative Systematic Bronchial Aspiration With Flexible Bronchoscope on Occurrence of Pulmonary Complications After Anatomical Lung Resections: a Prospective Randomized Controlled Study.
Brief Title: Influence of Postoperative Bronchoscopy on Pulmonary Complications After Anatomical Lung Resections.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wielkopolskie Centrum Pulmonologii i Torakochirurgii (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TH-17-BR-1
Record Dates: First submitted 2017-09-28; First posted 2017-10-11 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Postoperative Complications; Thoracic Surgery
Keywords: Bronchoscopy; Respiratory Complications; Anatomical Lung Resection
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bronch (Experimental): Postoperative systematic bronchial aspiration.
  Interventions: Procedure: Postoperative systematic bronchial aspiration.
- Control (No Intervention): In this arm bronchial aspiration with bronchoscope will not be done.

INTERVENTIONS:
Procedure: Postoperative systematic bronchial aspiration. — Postoperative flexible bronchoscopy and systematic bronchial aspiration.
  Arms: Bronch

SUMMARY:
Respiratory complications are the largest group of complications following anatomical lung resections. Most of these complications result from a disrupted evacuation of respiratory secretions. At present, prevention of such complications involve: aspirating of secretions with a catheter during surgery through an intubation tube, active postoperative rehabilitation, mucolytic treatment and effective postoperative pain management. Suctioning of secretions by a catheter through an intubation tube does not, however, allow for removal of secretions from entire bronchial tree. Bronchofiberoscopy with a small-diameter flexible bronchoscope and thorough, systematic aspiration of secretions from respiratory tract immediately after surgery could presumably result in more effective bronchial cleansing and reduce risk of respiratory complications after surgery. Although the British Thoracic Society guidelines do not recommend routine bronchoscopy as a standard postoperative management after lung resections, they are based on a single, randomized, study analyzing a small group of patients. Bronchoscopy with systematic aspiration of secretions done with a thin flexible scope is a safe procedure, without risk of complications. It does not cause any additional discomfort to the patients and allows for much more accurate aspiration of the bronchial secretions than with a catheter inserted blindly through an intubation tube. It also gives an opportunity to directly evaluate segmental and subsegmental bronchial patency. This is particularly important in patients with COPD who tend to accumulate large amounts of mucus secretion in the bronchial tree.

DETAILED DESCRIPTION:
Introduction.

Atelectasis and pneumonia are the most common complications after anatomical lung resections. Their occurrence in the postoperative period may necessitate treatment with antibiotics and fiberoptic bronchoscopy and may lead prolongation of hospital stay, diminished quality of life and increased cost of treatment.

Among known risk factors, retention of bronchial secretions is probably the most important. Although at the end of surgery suctioning of the secretions from large airways is always done, it is usually performed with suction catheter inserted blindly through an endotracheal tube. This procedure does not allow for complete removal of secretions from all parts of bronchial tree and trachea. Remaining secretions may lead to postoperative atelectasis and pneumonia.

Fiberoptic bronchoscopy performed with a thin scope allows for accurate visual assessment and precise aspiration of secretions from all main, lobar and segmental bronchi. If performed in a systematic way, it allows for complete removal of bronchial secretions.

The role of routine bronchoscopic aspiration has already been evaluated in one randomized study. However, study group included only 20 subjects, which is too little to perform proper statistical analysis and draw conclusions (1).

Study design.

After qualification for the study informed consent will be obtained from a patient.

Patients will be randomly assigned to one of two arms of the study: "BRONCH" or "CONTROL". Simple randomization method and random number generator (https://www.graphpad.com/quickcalcs/index.cfm) will be used.

Initial assessment will include demographics, smoking history, comorbidities (Charlson Comorbidity Index, CCI and Thoracic Revised Cardiac Risk Index, thRCRI), pulmonary function tests, diffusion lung capacity (DLCO), computed tomography of the chest and bronchoscopy.

Surgery will be performed under general anesthesia with double-lumen endotracheal tube intubation and single lung ventilation. Patients will be placed in lateral decubitus position and operation table will be flexed at the level of 5th - 6th rib The decision about the type of surgical approach (video-assisted thoracic surgery, VATS or antero-lateral muscle-sparing thoracotomy) will be made according to the criteria presently used, in particular size of a tumor and its TNM classification assessed on the basis of preoperative studies.

Pulmonary lobectomy will be performed in standardized fashion. Pulmonary vessels (veins and arteries) will be closed with vascular staplers, silk loops or vascular clips. Bronchus will be closed with stapler or running suture. Interlobar fissures will be divided with staplers. Mediastinal lymph node dissection (MLND) will be performed using either monopolar electrocautery or high-energy device. One chest tube will be placed in case of VATS and two in case of thoracotomy.

At the end of surgery, after lobectomy and MLND, catheter will be introduced through intubation tube and suctioning of secretions from large airways will be done. Collapsed lung will be re-expanded and alveolar recruitment maneuvers will be performed.

VATS/thoracotomy wound will be closed and patient will be placed in prone position. All investigators, except one designated for performing bronchoscopy will leave operating room.

At this time, it will be checked, to which arm the patient was randomly assigned. If the patient was assigned to "CONTROL" arm, bronchoscopy will not be done and the patient will be woken. If the patient was assigned to "BRONCH" arm, bronchoscopy will be done.

Bronchoscope will be kept in a closed cupboard, so it will not be possible for the investigators involved in perioperative assessment and surgery to accidentally learn if it has been used or not. If the patient will be assigned to "BRONCH" group, scope will be brought from the cupboard.

Bronchoscopy will be done with a thin, flexible bronchoscope by investigator specifically designated for the task, who will not participate in postoperative assessment of the patients. He/she will not be allowed to inform other investigators if bronchoscopy would be performed or not.

Bronchoscopy and suctioning of secretions will be performed in a systematic manner as follows: 1) main bronchi, 2) lung on non-operated side: lower lobe - middle lobe/lingula- upper lobe/culmen, 3) lung on operated side starting from lower lobe bronchi towards upper lobe bronchi, 4) main bronchi. Secretions will be removed from main, lobar and segmental bronchi. Care will be taken not to injure bronchial mucosa. Bronchial secretions will be sent for microbiological examination.

After bronchoscopy scope will be immediately transferred for cleaning and another one will be placed in the cupboard.

After operation patient will be transferred to surgery ward or intensive care unit if necessary.

Pain management will include local analgesia (epidural in thoracotomy, intercostal block with bupivacaine performed at the end of surgery in VATS), acetaminophen, NSAIDS and opioids. Pain severity will be assessed daily.

Physical examination, including auscultation, temperature measurement, heart rate, respiratory rate and others will be performed twice a day. Chest x-ray will be performed in the evening on the day of surgery, on postoperative day 1 and postoperative day 2 and additionally if symptoms corresponding to retention of secretions, atelectasis or pneumonia will be found on physical examination. C-reactive protein serum level will be measured before surgery and 72 hours after surgery.

The following factors/parameters will be additionally measured and compared in both groups: duration of surgery, duration of single-lung ventilation, chest tube duration, hospital stay, ICU admission and its duration, results of bacteriological examination of bronchial secretions, histology, TNM, stage.

Other complications will be recorded (bleeding, transfusion, prolonged air leak, residual air space, wound infection, redo surgery, psychosis and others).

Chest tubes will be removed if fluid drainage will be less than 200ml/day and no air leak will be observed.

Endpoints.

Primary endpoint:

1. Occurrence of atelectasis on chest x-ray on day 1, 2 or 3 after surgery

Secondary endpoint:

1. Bronchial Secretion Retention Related Complications Score (BRCS) on day 1, 2 or 3 after surgery
2. Occurrence of new atrial fibrillation during day 1, 2 or 3 after surgery
3. C-reactive protein level 72 hours after surgery

BRCS will reflect a spectrum of complications resulting from retention of bronchial secretions. Each of the complications will be assigned a number corresponding to severity of a complication (ordinal scale), as follows:

1. Normal breath sounds on auscultation, no atelectasis on CXR, no pneumonia.
2. Residual secretions on auscultation, no atelectasis on CXR, no pneumonia.
3. Atelectasis on CXR, no pneumonia.
4. Pneumonia.

Investigators plan to enroll 200 patients, 100 patients in each group.

Statistical analysis.

The analyzed data will be presented as means, standard deviations, minimum and maximum values, medians, interquartile ranges (lower quartile, upper quartile) or percentage, as appropriate. Normality of the distribution will be tested with the Shapiro-Wilk's test, and the equality of variances will be checked with the Levene's test. For comparison of groups, unpaired t test or one-way ANOVA (for data which follow normal distribution and homogeneity of variances) or Welch test will be applied. In case data will not normally distributed nonparametric tests will be used - Mann-Whitney U test or the Kruskal-Wallis test with the Dunn's post-hoc test. Categorical data will be analyzed with the χ2 test or the Fisher-Freeman-Halton test. The relationship between variables will be analyzed with the Pearson's linear correlation coefficient or the Spearman's rank correlation coefficient or (and) by multivariate linear regression. All the results will be considered significant at p<0.05. Statistical analyses will be performed with statistical packages: STATISTICA 10.0 PL (StatSoft. Inc.) or StatXact 9.0 (CytelStudio) software.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary lobectomy.
* Patients must be informed and must sign and give written informed consent.

Exclusion Criteria:

* Wedge resection, segmentectomy, pneumonectomy.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-04-08 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Atelectasis. | Up to 3 days after surgery.
  Occurrence of atelectasis on chest X-ray.

SECONDARY OUTCOMES:
Bronchial Secretion Retention Related Complications Score (BRCS). | Up to 3 days after surgery.
  BRCS will reflect a spectrum of complications resulting from retention of bronchial secretions. Each of the complication will be assigned a number in ordinal scale corresponding to severity of a complication, as follows:
  1. Normal breath sounds on auscultation, no atelectasis on CXR, no pneumonia.
  2. Residual secretions on auscultation, no atelectasis on CXR, no pneumonia.
  3. Atelectasis on CXR, no pneumonia.
  4. Pneumonia.
Atrial fibrillation. | Up to 3 days after surgery.
  Occurrence of new atrial fibrillation on physical examination confirmed by electrocardiography.
CRP. | 72 hours after the end of surgery.
  Serum C-reactive protein level

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Gabryel, MD, Principal Investigator — Wielkopolskie Centrum Pulmonologii i Torakochirurgii
Locations (1):
- Wielkopolskie Centrum Pulmonologii i Torakochirurgii, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jaworski A, Goldberg SK, Walkenstein MD, Wilson B, Lippmann ML. Utility of immediate postlobectomy fiberoptic bronchoscopy in preventing atelectasis. Chest. 1988 Jul;94(1):38-43. doi: 10.1378/chest.94.1.38. PMID 3289837
- [Background] Du Rand IA, Barber PV, Goldring J, Lewis RA, Mandal S, Munavvar M, Rintoul RC, Shah PL, Singh S, Slade MG, Woolley A; BTS Interventional Bronchoscopy Guideline Group. Summary of the British Thoracic Society guidelines for advanced diagnostic and therapeutic flexible bronchoscopy in adults. Thorax. 2011 Nov;66(11):1014-5. doi: 10.1136/thoraxjnl-2011-201052. PMID 22003155
- [Background] Stolz AJ, Schutzner J, Lischke R, Simonek J, Harustiak T, Pafko P. Predictors of atelectasis after pulmonary lobectomy. Surg Today. 2008;38(11):987-92. doi: 10.1007/s00595-008-3767-x. Epub 2008 Oct 29. PMID 18958555